CLINICAL TRIAL: NCT03054233
Title: Comparison of Successful Spinal Needle Insertion Between Obese and Non-obese Pregnant Women in Crossed Leg Sitting Position Undergoing Caesarean Section
Brief Title: Comparison of Successful Spinal Needle Insertion Between Obese and Non-obese Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Susilo Chandra, Anesthesiologist Consultant, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes010
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Caesarian Section
Keywords: spinal anesthesia; spinal-bone contact; caesarian section; crossed leg sitting position

ARMS (2):
- Obese (Experimental): Obese pregnant women received spinal anesthesia using Quincke Needle 25G/27G in crossed leg sitting position for caesarean section
  Interventions: Procedure: Crossed leg sitting position
- Non-obese (Experimental): Non-obese pregnant women received spinal anesthesia using Quincke Needle 25G/27G in crossed leg sitting position for caesarean section
  Interventions: Procedure: Crossed leg sitting position

INTERVENTIONS:
Procedure: Crossed leg sitting position — Spinal anesthesia done in crossed leg sitting position

SUMMARY:
The study aimed to compare successful spinal needle insertion between obese and non-obese pregnant women in crossed leg sitting position undergoing cesarean section

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine University of Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study.Subjects sat in cross leg sitting position: patients sit with both thighs abducted, knees flexed medially, each feet soles were under their contralateral thighs. The back was flexed maximally, subjects' chin approaching the sternum, and subjects hugged a pillow. Lumbal puncture was done using Quincke needle 25G/27G at L4-5 intervertebral gap until the it reached subarachnoid space (confirmed by free flow cerebrospinal fluid). Data recorded were the number of attempt for the successful spinal puncture, the number of spinal needle-bone contact and blood vessel puncture incidence. Data was analyzed by using Statistical Package for Social Scientist (SPSS), for numerical data using unpaired T-test or Mann-Whitney-U test, for categorical data using Chi-square test or Fischer Exact's Test. Data normality was tested by Kolmogorov-Smirnov test. Significant value is p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-45 years old, with American Society of Anesthesiologists (ASA) physical status I-III who were planned to undergo caesarian section with spinal anesthesia in crossed leg sitting position.
* Subjects have been explained about the study, have agreed to enroll and have signed the informed consent form

Exclusion Criteria:

* Subjects with contraindications for spinal anesthesia
* Subjects with fetal's head trapped, umbilical prolapse, and foot presentation
* Subjects with pre-eclampsia
* Subjects with cardiovascular diseases
* Subjects with scoliosis
* Subjects with recent lumbal surgery history
* Subjects who cannot sit in crossed leg sitting position.

Drop out criteria:

* Subjects with worsening conditions before spinal anesthesia
* Subjects with failed spinal needle insertion and thus received general anesthesia
* Subjects with twin pregnancy
* Subjects drop out the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of successful spinal needle placement in the first attempt | 2 months
  The number of successful spinal needle placement in the first attempt was recorded in yes/no method.
The number of needle-bone contact | 2 months
  The number of spinal needle-bone contact

SECONDARY OUTCOMES:
The number of blood vessel puncture incidence. | 2 months
  The number of blood vessel puncture incidence by the spinal needle during insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Susilo Chandra, Principal Investigator — Indonesia University
Locations (2):
- Indonesia (2):
  - Cipto Mangunkusumo Central National Hospital, Central Jakarta, DKI Jakarta
  - Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Davies GA, Maxwell C, McLeod L, Gagnon R, Basso M, Bos H, Delisle MF, Farine D, Hudon L, Menticoglou S, Mundle W, Murphy-Kaulbeck L, Ouellet A, Pressey T, Roggensack A, Leduc D, Ballerman C, Biringer A, Duperron L, Jones D, Lee LS, Shepherd D, Wilson K; Society of Obstetricians and Gynaecologists of Canada. SOGC Clinical Practice Guidelines: Obesity in pregnancy. No. 239, February 2010. Int J Gynaecol Obstet. 2010 Aug;110(2):167-73. doi: 10.1016/j.ijgo.2010.03.008. PMID 20641146
- [Background] American College of Obstetricians and Gynecologists. ACOG Committee opinion no. 549: obesity in pregnancy. Obstet Gynecol. 2013 Jan;121(1):213-7. doi: 10.1097/01.aog.0000425667.10377.60. PMID 23262963
- [Background] Rodrigues FR, Brandao MJ. Regional anesthesia for cesarean section in obese pregnant women: a retrospective study. Rev Bras Anestesiol. 2011 Jan-Feb;61(1):13-20. doi: 10.1016/S0034-7094(11)70002-2. PMID 21334503
- [Background] Soltani Mohammadi S, Hassani M, Marashi SM. Comparing the squatting position and traditional sitting position for ease of spinal needle placement: a randomized clinical trial. Anesth Pain Med. 2014 Apr 5;4(2):e13969. doi: 10.5812/aapm.13969. eCollection 2014 May. PMID 24790901
- [Background] Watanabe S, Kobara K, Ishida H, Eguchi A. Influence of trunk muscle co-contraction on spinal curvature during sitting cross-legged. Electromyogr Clin Neurophysiol. 2010 Apr-Jun;50(3-4):187-92. PMID 20552952
- [Background] Sebire NJ, Jolly M, Harris JP, Wadsworth J, Joffe M, Beard RW, Regan L, Robinson S. Maternal obesity and pregnancy outcome: a study of 287,213 pregnancies in London. Int J Obes Relat Metab Disord. 2001 Aug;25(8):1175-82. doi: 10.1038/sj.ijo.0801670. PMID 11477502
- [Background] Mhyre JM. Anesthetic management for the morbidly obese pregnant woman. Int Anesthesiol Clin. 2007 Winter;45(1):51-70. doi: 10.1097/AIA.0b013e31802b8a90. No abstract available. PMID 17215699
- [Background] Vricella LK, Louis JM, Mercer BM, Bolden N. Anesthesia complications during scheduled cesarean delivery for morbidly obese women. Am J Obstet Gynecol. 2010 Sep;203(3):276.e1-5. doi: 10.1016/j.ajog.2010.06.022. Epub 2010 Jul 31. PMID 20673866
- [Background] Broadbent CR, Maxwell WB, Ferrie R, Wilson DJ, Gawne-Cain M, Russell R. Ability of anaesthetists to identify a marked lumbar interspace. Anaesthesia. 2000 Nov;55(11):1122-6. doi: 10.1046/j.1365-2044.2000.01547-4.x. PMID 11069342
- [Background] Gulay U, Meltem T, Nadir SS, Aysin A. Ultrasound-guided evaluation of the lumbar subarachnoid space in lateral and sitting positions in pregnant patients to receive elective cesarean operation. Pak J Med Sci. 2015 Jan-Feb;31(1):76-81. doi: 10.12669/pjms.311.5647. PMID 25878618
- [Background] Kim SH, Kim DY, Han JI, Baik HJ, Park HS, Lee GY, Kim JH. Vertebral level of Tuffier's line measured by ultrasonography in parturients in the lateral decubitus position. Korean J Anesthesiol. 2014 Sep;67(3):181-5. doi: 10.4097/kjae.2014.67.3.181. Epub 2014 Sep 24. PMID 25302094
- [Background] Reinius H, Jonsson L, Gustafsson S, Sundbom M, Duvernoy O, Pelosi P, Hedenstierna G, Freden F. Prevention of atelectasis in morbidly obese patients during general anesthesia and paralysis: a computerized tomography study. Anesthesiology. 2009 Nov;111(5):979-87. doi: 10.1097/ALN.0b013e3181b87edb. PMID 19809292
- [Background] Collins JS, Lemmens HJ, Brodsky JB, Brock-Utne JG, Levitan RM. Laryngoscopy and morbid obesity: a comparison of the "sniff" and "ramped" positions. Obes Surg. 2004 Oct;14(9):1171-5. doi: 10.1381/0960892042386869. PMID 15527629
- [Background] Cadi P, Guenoun T, Journois D, Chevallier JM, Diehl JL, Safran D. Pressure-controlled ventilation improves oxygenation during laparoscopic obesity surgery compared with volume-controlled ventilation. Br J Anaesth. 2008 May;100(5):709-16. doi: 10.1093/bja/aen067. PMID 18407943
- [Background] McKay RE, Malhotra A, Cakmakkaya OS, Hall KT, McKay WR, Apfel CC. Effect of increased body mass index and anaesthetic duration on recovery of protective airway reflexes after sevoflurane vs desflurane. Br J Anaesth. 2010 Feb;104(2):175-82. doi: 10.1093/bja/aep374. Epub 2009 Dec 26. PMID 20037150
- [Background] Anuurad E, Shiwaku K, Nogi A, Kitajima K, Enkhmaa B, Shimono K, Yamane Y. The new BMI criteria for asians by the regional office for the western pacific region of WHO are suitable for screening of overweight to prevent metabolic syndrome in elder Japanese workers. J Occup Health. 2003 Nov;45(6):335-43. doi: 10.1539/joh.45.335. PMID 14676412